CLINICAL TRIAL: NCT05357885
Title: Quantitative SARS-CoV-2 Antibody Pre and Post Cardiopulmonary Bypass
Brief Title: Quantitative COVID-19 SARS-CoV-2 Antibody Pre and Post Cardiopulmonary Bypass
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Jordan Goldhammer, MD, Associate Professor, Thomas Jefferson University
Other Study IDs: 21D.1055
Record Dates: First submitted 2021-11-17; First posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Laboratory Assessment SARS-CoV-2 Antibody Levels Before and After Surgery for Patients Requiring Cardiopulmonary Bypass

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2 Antibody test — SARS-CoV-2 antibody test at Jefferson is Roche Elecsys Anti-SARS-CoV-2 immunoassays performed under FDA's Emergency Use Authorization.

SUMMARY:
This study is designed to compare the levels of SARS-CoV-2 antibody prior to cardiopulmonary bypass and after cardiopulmonary bypass (CPB).

DETAILED DESCRIPTION:
This study is designed to compare the levels of SARS-CoV-2 antibody prior to cardiopulmonary bypass and after cardiopulmonary bypass (CPB).

During CPB the patients' blood volume is removed from the body and sent through the CPB machine. CPB consists of a pump (to keep blood moving) and oxygenator (to oxygenate blood). The oxygenator or CPB circuitry may effect antibody levels. In addition, patients on CPB experience hemodilution from blood transfusion and priming volume from the CPB circuit. Hemodilution may effect antibody levels.

Prior to CPB, during standard of care lab drawn from standard of care arterial catheter, 0.5ml of plasma will be sent to the TJUH microbiology lab for Roche Elecsys Anti-SARS-CoV-2 immunoassay for pre-CPB quantitative antibody testing.

On morning of postoperative day 1, during standard of care lab draw from standard of care arterial catheter, 0.5ml of plasma will be sent to the TJUH microbiology lab for Roche Elecsys Anti-SARS-CoV-2 immunoassay for post-CPB quantitative antibody testing.

On morning of postoperative day 5, during standard of care lab draw, 0.5ml of plasma will be sent to the TJUH microbiology lab for Roche Elecsys Anti-SARS-CoV-2 immunoassay for post-CPB quantitative antibody testing. If patient is discharged from the hospital prior to postoperative day #5, this immunoassay will be omitted.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting for elective cardiac surgery with the use of cardiopulmonary bypass that have received 2 or 3 doses of FDA approved or Emergency Use Authorization Covid vaccine.

Exclusion Criteria:

* Age < 18.
* Patients with indeterminant history of vaccination schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting for elective cardiac surgery with the use of cardiopulmonary bypass that have received 2 or 3 doses of FDA approved or Emergency Use Authorization Covid vaccine
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
assess antibody levels before and after CPB. | preop and up to 5 days post op
  assess antibody levels before and after CPB.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States